CLINICAL TRIAL: NCT00366964
Title: Determine The Efficacy Of The Wavelight Mydon Laser For Hair Removal And Treatment of Leg Veins
Brief Title: The Efficacy Of The Wavelight Mydon Laser for Hair Removal And Treatment of Leg Veins
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 200412776-1
Record Dates: First submitted 2006-08-19; First posted 2006-08-22 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Leg Veins; Hair Removal
MeSH Terms: interventions — Laser Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Device (No Intervention)
  Interventions: Device: Laser Treatment; Device: Wave Light laser device for skin treatment

INTERVENTIONS:
Device: Laser Treatment — The laser treatment involves the use of an FDA approved laser device (510K Clearance certificate) for hair removal and treatment of leg veins for females having skin types III - VI. The pulses are of appropriate energy and pulse duration based on the skin type.
Device: Wave Light laser device for skin treatment — To determine efficacy of FDA approved Laser treatment for hair removal and leg veins. The Mydon Wavelight is a Long Pulsed Nd Yag Laser, Class IV 1064 nm 55W

SUMMARY:
This study is being done to compare the efficacy of an FDA cleared laser device with other similar systems in the market for the treatment of leg veins and hair removal in patients with darker skin type.

DETAILED DESCRIPTION:
The specific aim of the study is to determine the efficacy of this FDA approved laser for hair removal and treatment of leg veins in female patients having darker skin types (Fitzpatrick Skin type III-VI) and compare it with the efficacy of other similar commercial units available in the U.S.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients of Asian and darker skin type greater than or equal to 18 years of age.
2. Ability to give informed consent.

Exclusion Criteria:

1. Pregnancy.
2. Taking medications that are photosensitizing.
3. History of skin disease in the area to be treated over the last 6 months.
4. Ongoing cutaneous lupus erythematosus, morphea, alopecia areata, or severe folliculitis.
5. History of keloidal or hypertrophic scarring.
6. Have inadequate hair growth in the test area of axilla.
7. Have unrealistic expectations of the treatment.
8. Co-existing severe emotional, medical or surgical illness leading to the inability to meet the follow-up requirements.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2004-10; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Safety and efficacy of the treatment will determine the outcome. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel B Eisen, M.D., Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis Medical Center Department of Dermatology, Sacramento, California, United States

REFERENCES:
- See also: University of California-Davis Department of Dermatology Clinical Research — http://www.ucdmc.ucdavis.edu/dermatology/research/clinical